CLINICAL TRIAL: NCT04032405
Title: Clinical Evaluation of Injectable Platelet Rich Fibrin With Connective Tissue Graft for the Treatment of Deep Gingival Recession Defects. A Controlled Randomized Clinical Trial.
Brief Title: Clinical Evaluation of Injectable Platelet Rich Fibrin With Connective Tissue Graft for the Treatment of Deep Gingival Recession Defects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Mustafa Ozcan, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CukurovaU-PER
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Gingival Recession
Keywords: connective tissue graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF+CTG (Active Comparator): the combined connective tissue graft (CTG) with coronally advanced flap (CAF)
  Interventions: Procedure: CAF+CTG+i-prf
- CAF+CTG+i-prf (Experimental): the combined connective tissue graft (CTG) and injectable platelet rich fibrin (i-prf) with coronally advanced flap (CAF)
  Interventions: Procedure: CAF+CTG+i-prf

INTERVENTIONS:
Procedure: CAF+CTG+i-prf — combined connective tissue graft (CTG) and injectable platelet rich fibrin (i-prf) with coronally advanced flap (CAF)

SUMMARY:
Aim: The aim of this study was to determine whether the combined connective tissue graft (CTG) with injectable platelet rich fibrin (i-prf) with coronally advanced flap (CAF) improved root coverage of deep Miller Class I or II gingival recessions compared to CTG alone with CAF.

Methods: Seventy-two patients with Miller class I and II gingival recessions were enrolled. Thirty-six patients were randomly assigned to the test group (CAF+CTG+i-prf) or control group (CAF+CTG). Clinical evaluations were made at 6 months

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years of age,
* Periodontally and systemically healthy,
* FMPS and FMBS <15%,
* Presence of deep Miller class I and II gingival recession defect (≥3 mm in depth) at the buccal aspect of incisors,

Exclusion Criteria:

Smoking,

* Contraindications for surgery,
* Presence of recession defects associated with caries, deep abrasion, restoration or pulpal pathology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
gingival recession depth | six months
  the distance between the CEJ and gingival margin-measurements were performed at the midbuccal aspect of the teeth, by manual probe and were rounded up to the nearest millimetre
Keratized tissue height | six months
  measured from the mucogingival junction to the gingival margin-measurements were performed at the midbuccal aspect of the teeth, by manual probe and were rounded up to the nearest millimetre

CONTACTS AND LOCATIONS:
Overall Officials: onur ucak Turer, Study Director — CukurovaU Prof.
Locations (1):
- Cukurova University, Adana, Balcalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No